CLINICAL TRIAL: NCT05991518
Title: Phase Ib/II Clinical Study of IAH0968 in Combination With Gemcitabine and Cisplatin for the Treatment of HER2-Positive Unresectable Advanced/Metastatic Malignant Tumors and Cholangiocarcinoma
Brief Title: IAH0968 in Combination With GC for the Treatment of HER2-Positive Unresectable Advanced/Metastatic Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IAH0968-201
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: HER2 Gene Mutation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia - Dose escalation (Experimental): To determine the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and/or recommended phase II dose (RP2D) of intravenous IAH0968 in combination with the GC regimen for adult patients with HER2-positive advanced solid tumors who have failed standard treatment.
  Interventions: Combination Product: Injection of IAH0968+Gemcitabine+Cisplatin
- Phase IIa - Clinical Exploratory Stage (Experimental): The RP2D determined from the Phase Ib study is used as the first-line treatment for HER2-positive advanced or metastatic biliary tract cancer (BTC) patients who have not received prior systemic therapy. The efficacy of IAH0968 in combination with the GC regimen is compared to the efficacy of placebo in combination with the GC regimen based on the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, using the objective remission rate (ORR) as the evaluation criteria.
  Interventions: Combination Product: Injection of IAH0968+Gemcitabine+Cisplatin; Combination Product: Gemcitabine+Cisplatin

INTERVENTIONS:
Combination Product: Injection of IAH0968+Gemcitabine+Cisplatin — Administration of IAH0968 is given once per cycle, with each cycle defined as every 3 weeks.
  Other Names: IAH0968+GC
Combination Product: Gemcitabine+Cisplatin — Gemcitabine is administered at a dose of 1000 mg/m2 on the second day (D2) and ninth day (D9) of each cycle. At least 6 hours after the completion of gemcitabine infusion, cisplatin is administered at a dose of 70 mg/m2 on the second day (D2) of each cycle.
  Other Names: GC
  Arms: Phase IIa - Clinical Exploratory Stage

SUMMARY:
The study aims to evaluate the efficacy and safety of IAH0968 in combination with gemcitabine and cisplatin for the treatment of HER2-positive unresectable advanced/metastatic malignant tumors and cholangiocarcinoma. The study is divided into two stages: Phase Ib, an open-label, non-randomized, multicenter dose-escalation trial, and Phase II, a randomized, double-blind, parallel-controlled, multicenter trial.

DETAILED DESCRIPTION:
Phase Ib is an open-label, non-randomized, multicenter dose-escalation trial. It utilizes the classic "3+3" design to investigate the safety and tolerability of IAH0968 in combination with gemcitabine and cisplatin for the treatment of HER2-positive unresectable advanced/metastatic malignant tumors and cholangiocarcinoma.

Phase II study is a randomized, double-blind, parallel-controlled, multicenter research design. It aims to investigate the efficacy of IAH0968 in combination with gemcitabine and cisplatin for the treatment of HER2-positive unresectable advanced/metastatic malignant tumors and cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Phase Ib

1. The age of the participant should be 18 years or older.
2. The participant should have been diagnosed with HER2-positive advanced solid tumors that have failed standard treatment, as confirmed by pathological histology or cytology. Standard treatment failure is defined as disease progression during or after the last treatment, or inability to tolerate treatment due to severe toxicity (grade ≥ 4 hematologic toxicity or grade ≥ 3 non-hematologic toxicity following previous standard treatment). HER2 positivity is defined as proven HER2-positive through immunohistochemistry (IHC) staining and/or fluorescence in situ hybridization (FISH). The interpretation and standards for HER2 positivity in breast cancer will follow current breast cancer guidelines, and for HER2 positivity in cancers other than breast cancer, current gastric cancer guidelines will be followed (Appendix 9).
3. The GC regimen is the frontline standard treatment for the specific type of cancer (including urinary tract carcinoma, NSCLC, pancreatic cancer, nasopharyngeal carcinoma, etc.).
4. The participant should have at least one measurable lesion according to RECIST 1.1 criteria, and the measurable lesion should not have undergone any local treatment (including local radiotherapy, ablation, and intervention therapy).
5. The ECOG performance status should be 0 or 1 (refer to Appendix 3).
6. During the screening phase, the participant's organ functions should be relatively normal (upper limit of normal values based on the respective study center's range), including:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Hemoglobin (Hgb) ≥ 90 g/L
   * Platelet count (PLT) ≥ 90 × 109/L
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 × upper limit of normal (ULN), or ≤ 5.0 × ULN for patients with liver metastasis
   * Total bilirubin (TBIL) ≤ 1.5 × ULN
   * Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min calculated according to the Cockcroft-Gault formula (refer to Appendix 2)
   * All premenopausal women and women within 12 months of menopause should have a negative pregnancy test.
   * Left ventricular ejection fraction (LVEF) ≥ 50%.
   * Prothrombin time or international normalized ratio ≤ 1.5 × ULN, unless the patient is receiving anticoagulant therapy.

   If the patient has received platelet growth factors and/or granulocyte colony-stimulating factors prior to the above examinations, a washout period of at least 1 week is required.
7. The expected survival period should be ≥ 3 months.
8. The patient should agree to use at least one medically acceptable contraceptive method during the study treatment period and within 6 months following the end of the study treatment (for women: intrauterine device, oral contraceptives, or condoms, etc.; for men: condoms, abstinence, etc.), and female patients should not be lactating.

The patient should have full understanding of the study content, procedures, and potential risks and benefits, and should sign the informed consent form. The patient should demonstrate good compliance and be able to cooperate with the study and follow-up.

Phase IIa

1. The age of the participant should be 18 years or older.
2. The participant should have been diagnosed with locally advanced or metastatic HER2-positive BTC (biliary tract cancer) confirmed by pathological histology or cytology, and should not have received systemic chemotherapy treatment.
3. The participant should have at least one measurable lesion according to RECIST 1.1 criteria, and the measurable lesion should not have undergone any local treatment (including local radiotherapy, ablation, and intervention therapy).
4. The ECOG performance status should be 0 or 1 (refer to Appendix 3).
5. During the screening phase, the participant's organ functions should be relatively normal (upper limit of normal values based on the respective study center's range), including:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Hemoglobin (Hgb) ≥ 90 g/L
   * Platelet count (PLT) ≥ 90 × 109/L
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 × upper limit of normal (ULN), or ≤ 5.0 × ULN for patients with liver metastasis
   * Total bilirubin (TBIL) ≤ 1.5 × ULN
   * Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min calculated according to the Cockcroft-Gault formula (refer to Appendix 2)
   * All premenopausal women and women within 12 months of menopause should have a negative pregnancy test.
   * Left ventricular ejection fraction (LVEF) ≥ 50%.
   * Prothrombin time or international normalized ratio ≤ 1.5 × ULN, unless the patient is receiving anticoagulant therapy.
6. The expected survival period should be ≥ 3 months.
7. The patient should agree to use at least one medically acceptable contraceptive method during the study treatment period and within 6 months following the end of the study treatment (for women: intrauterine device, oral contraceptives, condoms, etc.; for men: condoms, abstinence, etc.), and female patients should not be lactating.

The patient should have full understanding of the study content, procedures, and potential risks and benefits, and should sign the informed consent form. The patient should demonstrate good compliance and be able to cooperate with the study and follow-up.

Exclusion Criteria:

Phase Ib

1. Known hypersensitivity reaction to any monoclonal antibody or a documented history of allergies to gemcitabine or cisplatin and its components.
2. Previous treatment: (1) Not recovered from adverse reactions caused by previous anti-tumor treatment to normal levels (according to CTCAE 5.0, hematologic toxicity ≥ Grade 2, non-hematologic toxicity ≥ Grade 1), excluding radiation-induced late toxicities considered irreversible by the investigator such as alopecia and skin pigmentation. (2) Patients who have received treatment with trastuzumab/pertuzumab and their biosimilars (mono-therapy, combination chemotherapy, ADC drugs, bispecific antibodies, etc.) within 4 weeks prior to enrollment. (3) Patients who have participated in other clinical trials within 4 weeks prior to enrollment and have used investigational drugs during this period. (4) Patients who have previously received GC regimen treatment for anti-tumor therapy and experienced relapse due to drug resistance.
3. Previous allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
4. Surgical procedures within 4 weeks prior to enrollment, and the investigator considers that the patient's condition has not recovered to a level allowing for initiation of this study treatment (excluding previous diagnostic biopsies and biliary stent placement/percutaneous transhepatic cholangiographic drainage procedures performed to relieve bile duct obstruction [PTBD]).
5. Vaccination with live vaccines within 4 weeks prior to enrollment, or receipt of blood transfusion within 2 weeks.
6. Radiotherapy other than focal palliative bone radiotherapy within 4 weeks prior to enrollment.
7. Clinical symptoms of central nervous system metastasis within 4 weeks prior to enrollment. Patients with previous treatment for brain or meningeal metastases may be included if the clinical condition is stable for at least 2 months and systemic steroid therapy (dose > 10 mg/day prednisone or equivalent) has been discontinued for ≥ 4 weeks.
8. Hospitalization or inability to undergo study treatment within 30 days prior to randomization due to exacerbation of chronic obstructive pulmonary disease or other respiratory diseases.
9. Liver transplant candidates and patients who can undergo transplantation during a medically acceptable period.
10. Exclusion of early-stage cancers (other than those treated with curative intent within 5 years before signing the informed consent), including but not limited to in situ cervical cancer, superficial noninvasive bladder cancer, basal cell carcinoma, and in situ squamous cell carcinoma, or gastrointestinal tumors limited to the mucosal layer and already resected under endoscopy.
11. Presence of severe or poorly controlled diseases, including but not limited to: (1) myocardial infarction, clinically significant arrhythmias requiring treatment, congestive heart failure, myocarditis, and angina pectoris occurring within 6 months prior to enrollment. (2) Hepatitis B virus (HBV) infection with positive HBV DNA (≥1.0×104 copies/mL or ≥2000 IU/mL), hepatitis C virus (HCV) infection with positive HCV RNA (>1.0×103 copies/mL or >100 IU/mL), and positive human immunodeficiency virus (HIV) test. (3) Active tuberculosis (clinical symptoms, physical examination findings, or radiographic evidence of active tuberculosis). (4) Severe and uncontrolled pulmonary diseases (severe infectious pneumonia, interstitial lung disease, etc.) (≥ Grade 3 CTCAE). (5) Uncontrolled biliary infection. Biliary obstruction should be relieved by endoscopic or percutaneous transhepatic biliary drainage (PTBD). Patients with biliary obstruction should have sufficient biliary drainage and no evidence of ongoing infection at the time of enrollment and on Day 1 of Cycle 1 without antibiotic treatment. (6) Severe infections of any type that are uncontrolled (≥ Grade 3 CTCAE). (7) Presence of ascites, pleural effusion, or pericardial effusion requiring drainage before the first study drug treatment.

Presence of other conditions considered inappropriate for participation in this study by the investigator.

Phase IIa

1. Known hypersensitivity reaction to any monoclonal antibody.
2. History of allergy to gemcitabine or cisplatin and its components.
3. Recent surgery within 4 weeks prior to enrollment, with the patient's condition considered inadequate for starting the study treatment (excluding prior diagnostic biopsies and percutaneous transhepatic biliary drainage PTBD for relieving bile duct obstruction).
4. Vaccination with any live vaccines within 4 weeks prior to enrollment or receipt of blood transfusion within 2 weeks.
5. Radiation therapy received within 4 weeks prior to enrollment, excluding focal palliative bone radiation.
6. Detection of clinically symptomatic central nervous system metastasis within 4 weeks prior to enrollment. Prior treatment for brain or meningeal metastasis is allowed if clinically stable for at least 2 months and has stopped systemic steroid therapy (dose >10 mg/day prednisone or equivalent) for ≥4 weeks.
7. Hospitalization or inability to initiate study treatment due to exacerbation of chronic obstructive pulmonary disease or other respiratory diseases within 30 days prior to randomization.
8. Liver transplant candidates and patients who are eligible for transplantation within a medically acceptable time frame.
9. Exclusion of early-stage cancers treated with curative intent within the past 5 years or mucosal cancers limited to gastroenteric mucosa and treated by endoscopic resection.
10. Presence of severe or poorly controlled diseases, including but not limited to: a) occurrence of myocardial infarction, clinically significant cardiac arrhythmias requiring treatment, congestive heart failure, myocarditis, or angina within 6 months prior to enrollment; b) Hepatitis B virus (HBV) infection with positive HBV DNA (≥1.0×104 copies/mL or ≥2000 IU/mL), hepatitis C virus (HCV) infection with positive HCV RNA (>1.0×103 copies/mL or >100 IU/mL), or positive human immunodeficiency virus (HIV) test; c) active tuberculosis (clinical symptoms, physical examination findings, or radiographic evidence of active tuberculosis); d) severe and uncontrolled pulmonary disease (severe infectious pneumonia, interstitial lung disease, etc.) (≥CTCAE Grade 3); e) uncontrolled biliary infection. Biliary obstruction should be relieved by stent placement or percutaneous transhepatic biliary drainage (PTBD). Patients with biliary obstruction should have adequate biliary drainage, with no evidence of ongoing infection on the day of enrollment and Day 1 of Cycle 1, without receiving antibiotic treatment; f) uncontrolled severe infections of any kind (≥CTCAE Grade 3); and g) presence of ascites, pleural effusion, or pericardial effusion requiring drainage prior to initial study drug treatment.

Other conditions deemed inappropriate for participation in this study, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Dose limiting toxicities (DLTs) (Phase Ⅰ) | 21 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
Objective response rate (ORR) in dose expansion (Phase Ⅱa) | Baseline through up to 1 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmax) following single dose.following single dose.
Pharmacokinetic (PK) Cmin (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmin) following single dose.following single dose.
Pharmacokinetic (PK) Tmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-t) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) CL (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CL) following single dose.
Pharmacokinetic (PK) Vd (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vd) following single dose.
Pharmacokinetic (PK) t1/2 (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,max) following multiple dose.
Pharmacokinetic (PK) Css,min (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,min) following multiple dose.
Pharmacokinetic (PK) Css,av (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,av) following multiple dose.
Pharmacokinetic (PK) AUCss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUCss) following multiple dose.
Pharmacokinetic (PK) CLss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CLss) following multiple dose.
Pharmacokinetic (PK) Vss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vss) following multiple dose.
Pharmacokinetic (PK) R (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (R) following multiple dose.
Pharmacokinetic (PK) DF (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (DF) following multiple dose.
Objective response rate (ORR) in dose escalation (Phase Ⅰ) | Baseline through up to 1 years or until disease progression
  Tumor response based on RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase Ⅰ) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAH0968.(Phase Ⅰb)
Progression free survival (PFS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1.
Overall survival (OS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
Disease control rate (DCR) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅱa) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase Ⅱa) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAH0968.(Phase Ⅱa)

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Jian, M.D., Principal Investigator — Fudan University; Liu Tianshu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Affiliated Zhongshan Hospital, Shanghai, China